CLINICAL TRIAL: NCT03659058
Title: Impact of Ursodeoxycholic Acid, Silymarin, Antioxidants and Colchicine on Fibrosis Regression in HCV After Achieving Sustained Virological Response
Brief Title: Impact of Ursodeoxycholic Acid, Silymarin, Antioxidants and Colchicine on Fibrosis Regression in HCV After SVR
Acronym: fib-reversal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor of medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37801
Record Dates: First submitted 2018-08-06; First posted 2018-09-06 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Fibrosis, Liver
Keywords: fibrosis; HCV; Reversal; sustained virological response
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Silymarin; Ursodeoxycholic Acid; Antioxidants; Colchicine; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: 200 patients will receive silymarin 420 mg + antioxidants + colchicine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): 200 patients with compensated liver cirrhosis (F4) by fibroscan; Child Turcotte Pugh score A, after achieving sustained virological response will be treated by anti-fibrotic agents
  Interventions: Drug: silymarin; Drug: Ursodeoxycholic Acid; Drug: Antioxidants; Drug: Colchicine; Other: FOLLOW UP
- control group (Placebo Comparator): 200 patients with compensated liver cirrhosis (F4) by fibroscan; Child Turcotte Pugh score A, after achieving sustained virological response will be followed up without any intervention
  Interventions: Other: FOLLOW UP

INTERVENTIONS:
Drug: silymarin — silymarin 140 three times daily
  Other Names: silymarin 140
  Arms: study group
Drug: Ursodeoxycholic Acid — Ursodeoxycholic Acid 500
  Other Names: ursofalk
  Arms: study group
Drug: Antioxidants — Beta Carotene - 6Mg Vitamin C - 200Mg Vitamin E - 50Mg
  Other Names: antox
  Arms: study group
Drug: Colchicine — Colchicine 0.6
  Arms: study group
Other: FOLLOW UP — follow up by abdominal ultrasound and fibroscan every 6 month for 1 year
  Other Names: ultrasound and fibroscan

SUMMARY:
with the introduction of Direct-acting antiviral agents in the management of HCV, the scope of inclusion criteria had been widened to include patients with compensated cirrhosis and even in special situations patients with decompensated liver disease; a chance that was not offered by the limited and strict inclusion criteria needed for treatment by pegylated interferon-based regimen. this made the number of patients with progressive liver fibrosis of cirrhosis had been inv=creased even after achieving SVR. the debate about the impact of SVR on halting fibrosis progression had risen; some studies postulated that patients benefit from an SVR through reduction of mortality, morbidity, and improved quality of life ; however, some patients may maintain their level of fibrosis or even progress to cirrhosis despite achieving SVR and the risk for HCC remains even after virologic eradication.

ELIGIBILITY:
Inclusion Criteria:

* chronic HCV
* compensated liver disease (Child class A-B)
* sustained virological response
* liver stiffness by fibroscan >12.5 kPa denotes cirrhosis

Exclusion Criteria:

* decompensated liver disease
* chronic active HCV
* hepatocellular carcinoma
* other liver diseases as alcoholic liver disease, autoimmune liver disease, drug-induced liver disease
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Improvement in liver stiffness measurement by Fibroscan | 1 year
  Liver stiffness assessment by Fibroscan every 6 months
Improved portal hypertension parameters | 1 year
  Assessment of portal vein diameter, splenic vein diameter, portal vein congestive index by ultrasound and Doppler every 6 months
Improved splenic stiffness measurement | 1 year
  assessment by ultrasound and fibroscan

IPD SHARING:
Plan to Share IPD: No